CLINICAL TRIAL: NCT00229879
Title: Rare Tumor Case Review
Status: Terminated | Type: Observational
Why Stopped: sufficient data gathered to support conclusion
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 04-119
Record Dates: First submitted 2005-09-13; First posted 2005-09-30 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2007-05

CONDITIONS: Intrapericardial Teratoma Tumor; Tumors
Keywords: pediatric health; rare tumor; children; cardiac
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to do a literature review and combine all of the cases of the intrapericardial teratoma tumor and see if some conclusions can be made about this rare tumor in children.

DETAILED DESCRIPTION:
We excised an intrapericardial teratoma tumor out of a child approximately one month ago.

This is a very uncommon tumor overall, and even more uncommon in children. The majority of reports in the literature are single case reports

I would like to report ours, as well as do a literature review to combine all of the cases and see if some conclusions can be made about this rare tumor in children.

ELIGIBILITY:
Inclusion Criteria:

* Children with intrapericardial teratoma tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with intrapericardial teratoma tumors
Sampling Method: Non-Probability Sample
Dates: Start 2004-12; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kogon, MD, Principal Investigator — Emory University; Kirk R Kanter, MD, Principal Investigator — Emory University; Paul M. Kirshbom, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States